CLINICAL TRIAL: NCT05554562
Title: Adductor Strength Assessment With Different Procedures for Athletes Suffering a Groin Injury
Brief Title: Adductor Strength in Athletes Suffering a Groin Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Principal Investigator, University of Oviedo
Other Study IDs: UO2022-04
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Groin Injury
Keywords: multidirectional sport; groin pain; adductor strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Injured athletes: Athletes suffering a groin injury
  Interventions: Other: Adductor strength assessment

INTERVENTIONS:
Other: Adductor strength assessment — Adductor strength will be evaluated with HHD (handheld dynamometer) and forceplates (Forceframe), both injured leg and healthy will be assess in order to compare both limbs

SUMMARY:
assess the difference in adductor peak strength evaluated with different instruments. Hand held dynamometer vs force frame

DETAILED DESCRIPTION:
This study aims to compare the difference in adductor strength output performed by athletes suffering a groin injury between two different assessment methods. Previous studies have observed that add strength differs depending on the evaluation method. Isometric strength can be measured with hand held dynamometer or with force plates (forceframe). Wether one method is better in order to differenciate adductor strength between healthy and injured limb is not known to date.

ELIGIBILITY:
Inclusion Criteria:

* Suffer a groin injury during the assessment period
* Accept participating in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: athletes from multidirectional sports (football, basketball, hockey, etc) currently suffering a groin injury
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
handheld dynamometer strength | november 2022 to june 2023
  peak torque measured with the handheld dynamometer the athlete will lay supine with hips flexed at 0º and the examiner will put the forearm between the ankles, the participant has to exert the maximum possible strength with the adductor muscles by squeezing with both legs against the forearm
forceframe strength | november 2022 to june 2023
  peak torque measured with the forceframe the athlete will lay supine with hips flexed at 0º and the ankles placed by the force plates, the participant has to exert the maximum possible strength with the adductor muscles by squeezing with both legs against the plates

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Olmedillas, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No